CLINICAL TRIAL: NCT06515197
Title: Investigating the Effects of Music on Mental Energy, Mental Toughness, Psychological Skills, Mindfulness, Athletic Identity, and Sports Performance Among Young Basketball Players
Brief Title: Effects of Music on Mental and Physical Performance in Young Basketball Players
Acronym: MEPMSAP-YBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, SHUAI YING, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MEPMSAP-YBP
Record Dates: First submitted 2024-07-09; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Mental Energy; Sports Performance; Basketball; Music Therapy; Adolescent Health; Mindfulness
Keywords: Music intervention; sports performance; adolescent basketball player; mental and physical health

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment model with three arms: motivational music, self-selected music, and no music control.
Masking Description: No masking is used in this study as participants and investigators are aware of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational Music (Experimental): Participants in this group will listen to pre-selected motivational music tracks for 30 minutes before each basketball training and performance test. This intervention will be conducted three times a week for 12 weeks. The aim is to assess the impact of motivational music on mental energy, mental toughness, psychological skills, mindfulness, athletic identity, and sports performance.
  Interventions: Other: Motivational Music
- Self-Selected Music (Experimental): Participants in this group will choose their own music to listen to for 30 minutes before each basketball training and performance test. This intervention will be conducted three times a week for 12 weeks. The goal is to determine the effect of self-selected music on mental energy, mental toughness, psychological skills, mindfulness, athletic identity, and sports performance.
  Interventions: Other: Self-Selected Music
- No Music Control (No Intervention): Participants in this group will not listen to any music before basketball training and performance tests. This control group will help compare the effects of no music intervention against the motivational and self-selected music interventions. The sessions will be conducted three times a week for 12 weeks.

INTERVENTIONS:
Other: Motivational Music — Participants in this group will listen to pre-selected motivational music tracks for 30 minutes before each basketball training and performance test. This intervention will be conducted three times a week for 12 weeks. The aim is to assess the impact of motivational music on mental energy, mental toughness, psychological skills, mindfulness, athletic identity, and sports performance.
  Arms: Motivational Music
Other: Self-Selected Music — Participants in this group will choose their own music to listen to for 30 minutes before each basketball training and performance test. This intervention will be conducted three times a week for 12 weeks. The goal is to determine the effect of self-selected music on mental energy, mental toughness, psychological skills, mindfulness, athletic identity, and sports performance.
  Arms: Self-Selected Music

SUMMARY:
The goal of this clinical trial is to evaluate if different music interventions (motivational music, self-selected music, and no music) can enhance mental and physical performance in young basketball players aged 12-19 in Shandong Province, China. The primary questions it aims to answer are:

Does motivational music lead to higher levels of mental energy, mental toughness, mindful attention awareness, psychological skills, and athletic identity compared to no music? Does self-selected music lead to higher levels of these variables compared to no music? Researchers will compare three groups (motivational music, self-selected music, and no music) to determine if these interventions significantly affect mental energy, mental toughness, psychological skills, mindfulness, athletic identity, and sports performance.

Participants will:

Be randomly assigned to one of three groups: motivational music, self-selected music, or no music (control).

Listen to their assigned type of music for 30 minutes before basketball training and performance tests, three times a week for 12 weeks.

Complete questionnaires and performance tests at the start and end of the study to measure changes in their mental and physical performance.

DETAILED DESCRIPTION:
Study Title:

Investigating the Effects of Music on Mental Energy, Mental Toughness, Psychological Skills, Mindfulness, Athletic Identity, and Sports Performance among Young Basketball Players in Shandong Province, China

Objective:

The objective of this clinical trial is to explore how different types of music (motivational, self-selected, and no music) affect the mental and physical performance of young basketball players aged 12-19 in Shandong Province, China.

Study Design:

This study is a single-center interventional randomized controlled trial with parallel assignment. It involves three groups: motivational music, self-selected music, and no music (control). There is no masking in this study.

Study Setting:

The study is conducted at a sports training center in Shandong Province, China.

Interventions:Participants are randomly assigned to one of three groups:

Motivational Music Group: Listens to pre-selected motivational tracks Self-Selected Music Group: Chooses their own music Control Group: Does not listen to any music Each group consists of 14 young basketball players. The intervention involves listening to the assigned type of music for a duration of 30 minutes before engaging in basketball training and performance tests, conducted three times a week for eight weeks.

Outcome Measures:Primary Outcome Measures: Mental Energy: Measured using the Athletic Mental Energy Scale (AMES) at pre-intervention and post-intervention (after 12 weeks).

Psychological Skills: Measured using the Psychological Skills Inventory (APSI) at pre-intervention and post-intervention (after 12 weeks).

Athletic Identity: Measured using the Athletic Identity Measurement Scale - Plus (AIMS-P) at pre-intervention and post-intervention (after 12 weeks).

Mindfulness: Measured using the Mindfulness Attention Awareness Scale (MAAS) at pre-intervention and post-intervention (after 12 weeks).

Mental Toughness: Measured using the Trait Mental Toughness Inventory for Sport (TMTIS) at pre-intervention and post-intervention (after 12 weeks).

Sport Performance Success: Measured using the Sport Success Scale (SSS) at pre-intervention and post-intervention (after 12 weeks).

Secondary Outcome Measures: Sports Performance: Measured through multiple crossover dribble layup, running vertical jump, and shooting tests at pre-intervention and post-intervention (after 12 weeks).

Hypotheses:

1. The level of mental energy, mental toughness, mindful attention awareness, psychological skills, athletic identity, and sports performance can be reliably measured using the AMES, MAAS, TMTIS, APSI, AIMS-P, and SSS scales, with average or total scores representing each domain.
2. Music intervention (motivational, self-selected, and no music) will have significant effects on mental energy, mental toughness, mindful attention awareness, psychological skills, and athletic identity among young basketball players.

   Motivational music will lead to higher levels of these variables compared to no music.

   Self-selected music will lead to higher levels of these variables compared to no music.
3. Music intervention will significantly affect sports performance. Motivational music will enhance sports performance more than no music. Self-selected music will enhance sports performance more than no music.

ELIGIBILITY:
Inclusion Criteria:

Youth basketball players with Chinese nationality Aged 15-17 years old Able to complete the questionnaires before and after the intervention Members of the same team with identical weekly training frequency, diet, and routine before and after the intervention At least 2 years of training experience No recent competition commitments Statistically insignificant differences in height, weight, and BMI

Exclusion Criteria:

Unwillingness to participate in the intervention phase Disabilities preventing physical activity Potential injuries or medical problems that could compromise participation or performance in the study

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Mental Energy | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Description: Mental energy will be measured using the Athletic Mental Energy Scale (AMES).
  Scale Title: Athletic Mental Energy Scale (AMES) Minimum and Maximum Values: The AMES ranges from 1 to 6. Score Interpretation: Higher scores indicate higher levels of mental energy. Time Frame: Baseline (pre-intervention) and 12 weeks (post-intervention).
Psychological Skills | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Description: Psychological skills will be measured using the Athletic Psychological Skills Inventory (APSI).
  Scale Title: Athletic Psychological Skills Inventory (APSI) Minimum and Maximum Values: The APSI ranges from 1 to 5. Score Interpretation: Higher scores indicate better psychological skills.
Athletic Identity | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Description: Athletic identity will be measured using the Athletic Identity Measurement Scale - Plus (AIMS-P).
  Scale Title: Athletic Identity Measurement Scale - Plus (AIMS-P) Minimum and Maximum Values: The AIMS-P ranges from 1 to 11. Score Interpretation: Higher scores indicate a stronger athletic identity.
Mindfulness | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Description: Mindfulness will be measured using the Mindfulness Attention Awareness Scale (MAAS).
  Scale Title: Mindfulness Attention Awareness Scale (MAAS) Minimum and Maximum Values: The MAAS ranges from 1 to 6. Score Interpretation: Higher scores indicate greater mindfulness.
Mental Toughness | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Description: Mental toughness will be measured using the Trait Mental Toughness Inventory for Sport (TMTIS).
  Scale Title: Trait Mental Toughness Inventory for Sport (TMTIS) Minimum and Maximum Values: The TMTIS ranges from 1 to 5. Score Interpretation: Higher scores indicate greater mental toughness.
Sports Performance Tests | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Description: Sports performance will be assessed through multiple tests including crossover dribble layup, running vertical jump, and shooting tests.
  Specific Tests:
  Crossover Dribble Layup Test: Number of successful layups in a given time frame.
  Running Vertical Jump Test: Height of vertical jump in centimeters. Shooting Test: Number of successful shots made in a given number of attempts.

CONTACTS AND LOCATIONS:
Locations (1):
- Shuai Ying, Rizhao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study will be available upon request from PhD candidate . The type of data to be shared includes individual participant data (IPD) such as responses to AMES, MAAS, TMTIS, APSI, AIMS-P, SSS questionnaires, and results from basketball performance tests. Data will become available six months after the study's results are published and will remain available for five years following publication. Access to the data will be granted to researchers who provide a methodologically sound proposal, subject to review and approval by the study team. Data will be anonymized to protect participant confidentiality. Researchers requesting data will need to sign a data access agreement.
Supporting Information: Study Protocol, ICF
Time Frame: The datasets generated during and/or analyzed during the current study will be available upon request from PhD candidate . The type of data to be shared includes individual participant data (IPD) such as responses to AMES, MAAS, TMTIS, APSI, AIMS-P, SSS questionnaires, and results from basketball performance tests. Data will become available six months after the study's results are published and will remain available for five years following publication. Access to the data will be granted to researchers who provide a methodologically sound proposal, subject to review and approval by the study team. Data will be anonymized to protect participant confidentiality. Researchers requesting data will need to sign a data access agreement.
Access Criteria: The datasets generated during and/or analyzed during the current study will be available upon request from PhD candidate . The type of data to be shared includes individual participant data (IPD) such as responses to AMES, MAAS, TMTIS, APSI, AIMS-P, SSS questionnaires, and results from basketball performance tests. Data will become available six months after the study's results are published and will remain available for five years following publication. Access to the data will be granted to researchers who provide a methodologically sound proposal, subject to review and approval by the study team. Data will be anonymized to protect participant confidentiality. Researchers requesting data will need to sign a data access agreement.

REFERENCES:
- [Background] Elliott D, Polman R, Taylor J. The effects of relaxing music for anxiety control on competitive sport anxiety. Eur J Sport Sci. 2014;14 Suppl 1:S296-301. doi: 10.1080/17461391.2012.693952. Epub 2012 Jun 19. PMID 24444221
- [Background] Priest DL, Karageorghis CI, Sharp NC. The characteristics and effects of motivational music in exercise settings: the possible influence of gender, age, frequency of attendance, and time of attendance. J Sports Med Phys Fitness. 2004 Mar;44(1):77-86. PMID 15181394
- [Result] Terry PC, Karageorghis CI, Curran ML, Martin OV, Parsons-Smith RL. Effects of music in exercise and sport: A meta-analytic review. Psychol Bull. 2020 Feb;146(2):91-117. doi: 10.1037/bul0000216. Epub 2019 Dec 5. PMID 31804098

DOCUMENTS (2):
  • Study Protocol (2022-10-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT06515197/Prot_000.pdf
  • Informed Consent Form (2022-10-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT06515197/ICF_001.pdf